CLINICAL TRIAL: NCT03251378
Title: A Multi-Center, Open-Label, Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Anticancer Activity of Fruquintinib in Patients With Advanced Solid Tumors
Brief Title: A Multi-Center, Open-Label Study of Fruquintinib in Solid Tumors and Colorectal, and Breast Cancers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hutchison Medipharma Limited (Industry)
Responsible Party: Sponsor
Organization: Hutchmed (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2015-013-00US1
Record Dates: First submitted 2017-07-19; First posted 2017-08-16 (Actual); Results first posted 2024-09-25 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-05

CONDITIONS: Advanced Solid Tumors; Metastatic Colon Cancer; Metastatic Breast Cancer; Triple Negative Breast Cancer; HER2-negative Breast Cancer; Hormone Receptor Positive Breast Carcinoma; Rectal Cancer
Keywords: VEGF; colorectal; breast
MeSH Terms: conditions — Colonic Neoplasms; Breast Neoplasms; Triple Negative Breast Neoplasms; Rectal Neoplasms | interventions — HMPL-013

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- 3 mg Dose Escalation (Experimental): 3 mg of Fruquintinib (HMPL-013), capsule taken orally, daily, 3 weeks on, 1 week off
  Interventions: Drug: Fruquintinib (HMPL-013)
- 5 mg Dose Escalation (Experimental): 5 mg of Fruquintinib (HMPL-013), capsule taken orally, daily, 3 weeks on, 1 week off
  Interventions: Drug: Fruquintinib (HMPL-013)
- Fruquintinib Expansion Cohort A (Experimental): 5 mg fruquintinib (HMPL-013) capsule taken orally, daily, 3 weeks on, 1 week off in patients with advanced solid tumors of any type.
  Interventions: Drug: Fruquintinib (HMPL-013)
- Metastatic Colorectal Cancer Expansion Cohort B (prior trifluridine/tipiracil or regorafenib) (Experimental): 5 mg fruquintinib (HMPL-013) capsule taken orally, daily, 3 weeks on, 1 week off in patients with metastatic colorectal cancer who have progressed on or had intolerable toxicity to TAS-102, regoragenib, or both.
  Interventions: Drug: Fruquintinib (HMPL-013)
- Metastatic Colorectal Cancer Expansion Cohort C (no prior trifluridine/tipiracil or regorafenib) (Experimental): 5 mg fruquintinib (HMPL-013) capsule taken orally, daily, 3 weeks on, 1 week off in patients with metastatic colorectal cancer who have not been treated with TAS-102 or regorafenib.
  Interventions: Drug: Fruquintinib (HMPL-013)
- Metastatic Breast Cancer (HR positive, HER2 negative) Expansion Cohort D (Experimental): 5 mg fruquintinib (HMPL-013) capsule taken orally, daily, 3 weeks on, 1 week off in patients with metastatic Her2-negative, hormone receptor positive breast cancer.
  Interventions: Drug: Fruquintinib (HMPL-013)
- Metastatic Breast Cancer (TNBC) Expansion Cohort E (Experimental): 5 mg fruquintinib (HMPL-013) capsule taken orally, daily, 3 weeks on, 1 week off in patients with metastatic triple negative (Her2-negative, ER-negative, PR-negative) breast cancer.
  Interventions: Drug: Fruquintinib (HMPL-013)

INTERVENTIONS:
Drug: Fruquintinib (HMPL-013) — Fruquintinib is a small molecule tyrosine kinase inhibitor (TKI) that targets VEGFR-1, -2, and -3, with a novel chemical structure which belongs to the quinazoline class.
  Other Names: HMPL-013

SUMMARY:
An open-label, dose escalation and expansion clinical trial to evaluate the safety, tolerability, and PK of fruquintinib in patients with advanced solid tumors, metastatic colorectal cancer and metastatic breast cancer.

DETAILED DESCRIPTION:
The study was an open-label, dose escalation and expansion clinical trial to evaluate the safety, tolerability, and PK of fruquintinib in patients with advanced solid tumors. The study consisted of two phases:

* A dose escalation phase - Two dose cohorts were evaluated including 3 mg orally QD 3 weeks on/1 week off and 5 mg orally QD 3 weeks on/1 week off. A 3+3 design was used for this portion of the study.
* A dose expansion phase - Five cohorts were evaluated in Dose Expansion phase. Cohort A evaluated the MTD/RP2D in patients with advanced solid tumors of any type. Cohort B and Cohort C evaluated the MTD/RP2D in metastatic colorectal cancer patients. Cohort D and Cohort E evaluated the MTD/RP2D in metastatic breast cancer patients.

Study was conducted at 9 sites in the United States.

ELIGIBILITY:
Key Inclusion Criteria:

* Fully understand the study and voluntarily sign the ICF;
* ≥18years of age;
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1;

Dose Escalation Phase:

• Histologically or cytologically documented, locally advanced or metastatic solid malignancy of any type (except squamous NSCLC) that has progressed on approved systemic therapy, and for whom no effective therapy or standard of care exists. This cohort is closed to enrollment.

Dose Expansion Phase:

* Cohort A: Histologically or cytologically documented, locally advanced or metastatic solid malignancy of any type (except squamous NSCLC), that has progressed on approved systemic therapy, and for whom no effective therapy or standard of care exists. This cohort is closed to enrollment.
* Cohort B: Histologically or cytologically documented mCRC in patients that have progressed on, or had intolerable toxicity with at least 1 FDA-approved third-line systemic therapy (trifluridine/tipiracil or regorafenib). Patients must also have been previously treated with fluoropyrimidine-, oxaliplatin-, and irinotecan-based chemotherapy, an anti-VEGF biological therapy, and an anti-EGFR therapy for patients who had RAS wild-type tumors. This cohort is currently enrolling.
* Cohort C: Histologically or cytologically documented adenocarcinoma of the colon or rectum. Patients must have progressed on, or had intolerable toxicity to, at least 2 prior regimens of standard chemotherapy, but must not have received prior TAS-102 or regorafenib. Prior therapy could have included adjuvant chemotherapy if a tumor had recurred within 6 months after the last administration of treatment. Patients must have been previously treated with fluoropyrimidine-, oxaliplatin-, and irinotecan-based chemotherapy, an anti-VEGF biological therapy and, if RAS wild-type, an anti-EGFR therapy
* Cohort D only: Histologically- or cytologically-confirmed Her2-negative, hormone receptor positive (ER+ and/or PR+) breast cancer
* Cohort E only: Histologically- or cytologically- confirmed triple negative breast cancer

Key Exclusion Criteria:

Patients will be excluded from the study, if any of the following criteria is met:

* Severe anemia, neutropenia, thrombocytopenia
* Moderate to severe renal or hepatic impairment
* Uncontrolled hypertension
* Risk of, or active hemorrhage: history or presence of active gastric/duodenal ulcer or ulcerative colitis, active hemorrhage of an unresected gastrointestinal tumor, history of perforation of fistulas; or any other condition that could possibly result in gastrointestinal tract hemorrhage or perforation within 6 months prior to screening;
* History of a thromboembolic event (including deep vein thrombosis [DVT], pulmonary embolism, stroke and/or transient ischemic attack) within 6 months prior to screening;
* Patients with squamous NSCLC;
* Clinically significant cardiovascular disease, including but not limited to acute myocardial infarction or coronary artery bypass surgery within 6 months prior to enrollment, severe or unstable angina pectoris, New York Heart Association Class III/IV congestive heart failure, ventricular arrhythmias requiring treatment, or left ventricular ejection fraction (LVEF) <50%;
* Patients who have ever received a VEGFR inhibitor, except for patients with mCRC enrolled in the dose expansion phase;
* Systemic anti-neoplastic therapies or any investigational therapy within 4 weeks prior to the first dose of study drug, including chemotherapy, radical radiotherapy, hormonotherapy, biotherapy and immunotherapy;
* Systemic small molecule targeted therapies (e.g., tyrosine kinase inhibitors) within 5 half-lives or 4 weeks (whichever is shorter) prior to the first dose of study drug;
* Palliative radiotherapy for bone metastasis/lesion within 2 weeks prior to the initiation of study drug;
* Brachytherapy (ie, implantation of radioactive seeds) within 60 days prior to the first dose of study drug;
* Known human immunodeficiency virus (HIV) infection;
* Known clinically significant history of liver disease, including cirrhosis, current alcohol abuse or active viral hepatitis. For patients with evidence of chronic hepatitis B (HBV), the HBV viral load must be undetectable on suppressive therapy, if indicated. Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV who are currently on treatment, they are eligible if they have an undetectable HCV viral load;
* Tumor invasion of a large vascular structure, eg, pulmonary artery, superior or inferior vena cava.;
* Women who are pregnant or lactating;
* Brain metastases and/or spinal cord compression untreated with surgery and/or radiotherapy, and without clinical imaging evidence of stable disease for 14 days or longer; patients requiring steroids within 4 weeks prior to start of study treatment will be excluded;
* No other malignancy, except for non-melanoma skin cancer, during the 5 years prior to screening;
* Inability to take medication orally, dysphagia or an active gastric ulcer resulting from previous surgery (eg, gastric bypass) or a severe gastrointestinal disease, or any other condition that investigators believe may affect absorption of the investigational product;
* Other disease, metabolic disorder, physical examination anomaly, abnormal laboratory result, or any other condition that investigators suspect may prohibit use of the investigational product, affect interpretation of study results, or put the patient at undue risk of harm based on the investigator's assessment;
* Known hypersensitivity to fruquintinib or any of its excipients.
* For Cohort C only: patients who have been previously treated with TAS-102 or regorafenib

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2017-12-11 (Actual); Primary Completion 2022-12-13 (Actual); Study Completion 2023-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Schelman, Study Director — HUTCHMED International
Locations (9):
- United States (9):
  - Mayo Clinic Arizona, Phoenix, Arizona
  - California Cancer Care Associates for Research & Excellence, Inc., San Marcos, California
  - St. Joseph Heritage Healthcare, Santa Rosa, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - Hem-Onc Associates of the Treasure Coast, Port Saint Lucie, Florida
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Vanderbilt Ingram Cancer Center, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang-Gillam A, Schelman W, Ukrainskyj S, Chien C, Gonzalez M, Yang Z, Kania M, Yeckes-Rodin H. Phase 1/1b open-label, dose-escalation study of fruquintinib in patients with advanced solid tumors in the United States. Invest New Drugs. 2023 Dec;41(6):851-860. doi: 10.1007/s10637-023-01395-y. Epub 2023 Oct 5. PMID 37796398

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 9 study sites in the United States.
Pre-assignment Details: A total of 129 participants (14 in Dose Escalation Phase and 115 in Dose Expansion Phase) were treated in this study.
Groups:
- Dose Escalation Phase: Fruquintinib 3 mg: Participants with advanced solid tumors of any type received fruquintinib 3 milligram (mg) capsules (3 capsules, 1mg/capsule), once daily, 3 weeks on, 1 week off in each 28-day treatment cycle until disease progression, unacceptable toxicity, use of other antitumor treatment, withdrawal of consent, or discontinuation by Investigator, whichever occurred first.
- Dose Escalation Phase: Fruquintinib 5 mg; Dose Expansion Phase, Cohort A: Fruquintinib 5 mg: Participants with advanced solid tumors of any type received fruquintinib 5 mg capsule, once daily, 3 weeks on, 1 week off in each 28-day treatment cycle until disease progression, unacceptable toxicity, use of other antitumor treatment, withdrawal of consent, or discontinuation by Investigator, whichever occurred first.
- Dose Expansion Phase, Cohort B: Fruquintinib 5 mg: Participants with metastatic colorectal carcinoma (mCRC) and prior treatment with trifluridine, tipiracil or regorafenib received fruquintinib 5 mg capsule, once daily, 3 weeks on, 1 week off in each 28-day treatment cycle until disease progression, unacceptable toxicity, use of other antitumor treatment, withdrawal of consent, or discontinuation by Investigator, whichever occurred first.
- Dose Expansion Phase, Cohort C: Fruquintinib 5 mg: Participants with mCRC and no prior treatment with trifluridine, tipiracil or regorafenib received fruquintinib 5 mg capsule, once daily, 3 weeks on, 1 week off in each 28-day treatment cycle until disease progression, unacceptable toxicity, use of other antitumor treatment, withdrawal of consent, or discontinuation by Investigator, whichever occurred first.
- Dose Expansion Phase, Cohort D: Fruquintinib 5 mg: Participants with hormone-receptor-positive (HR+), human epidermal growth factor receptor 2 (HER2)-negative metastatic breast cancer (mBC) received fruquintinib 5 mg capsule, once daily, 3 weeks on, 1 week off in each 28-day treatment cycle until disease progression, unacceptable toxicity, use of other antitumor treatment, withdrawal of consent, or discontinuation by Investigator, whichever occurred first.
- Dose Expansion Phase, Cohort E: Fruquintinib 5 mg: Participants with triple negative breast cancer (TNBC) received fruquintinib 5 mg capsule, once daily, 3 weeks on, 1 week off in each 28-day treatment cycle until disease progression, unacceptable toxicity, use of other antitumor treatment, withdrawal of consent, or discontinuation by Investigator, whichever occurred first.
Period: Overall Study
Arm/Group | Dose Escalation Phase: Fruquintinib 3 mg | Dose Escalation Phase: Fruquintinib 5 mg | Dose Expansion Phase, Cohort A: Fruquintinib 5 mg | Dose Expansion Phase, Cohort B: Fruquintinib 5 mg | Dose Expansion Phase, Cohort C: Fruquintinib 5 mg | Dose Expansion Phase, Cohort D: Fruquintinib 5 mg | Dose Expansion Phase, Cohort E: Fruquintinib 5 mg
Started | 7 | 7 | 6 | 41 | 40 | 14 | 14
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 7 | 7 | 6 | 41 | 40 | 14 | 14
Not completed — Death | 3 | 2 | 3 | 30 | 24 | 12 | 12
Not completed — Lost to Follow-up | 0 | 0 | 1 | 3 | 0 | 0 | 0
Not completed — Patient withdrew consent and refused to provide follow-up information | 0 | 0 | 0 | 3 | 2 | 1 | 1
Not completed — Progressive disease | 2 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 2 | 3 | 2 | 0 | 1 | 1 | 1
Not completed — Other | 0 | 0 | 0 | 4 | 13 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The safety analysis set (SAS) included all participants who received at least 1 dose of the study drug.
Groups:
- Dose Escalation Phase: Fruquintinib 3 mg: Participants with advanced solid tumors of any type received fruquintinib 3 mg capsules (3 capsules, 1mg/capsule), once daily, 3 weeks on, 1 week off in each 28-day treatment cycle until disease progression, unacceptable toxicity, use of other antitumor treatment, withdrawal of consent, or discontinuation by Investigator, whichever occurred first.
- Dose Expansion Phase, Cohort B: Fruquintinib 5 mg: Participants with mCRC and prior treatment with trifluridine, tipiracil or regorafenib received fruquintinib 5 mg capsule, once daily, 3 weeks on, 1 week off in each 28-day treatment cycle until disease progression, unacceptable toxicity, use of other antitumor treatment, withdrawal of consent, or discontinuation by Investigator, whichever occurred first.
- Dose Expansion Phase, Cohort D: Fruquintinib 5 mg: Participants with HR+, HER2-negative mBC received fruquintinib 5 mg capsule, once daily, 3 weeks on, 1 week off in each 28-day treatment cycle until disease progression, unacceptable toxicity, use of other antitumor treatment, withdrawal of consent, or discontinuation by Investigator, whichever occurred first.
- Dose Expansion Phase, Cohort E: Fruquintinib 5 mg: Participants with TNBC received fruquintinib 5 mg capsule, once daily, 3 weeks on, 1 week off in each 28-day treatment cycle until disease progression, unacceptable toxicity, use of other antitumor treatment, withdrawal of consent, or discontinuation by Investigator, whichever occurred first.
- Total: Total of all reporting groups
Arm/Group | Dose Escalation Phase: Fruquintinib 3 mg | Dose Escalation Phase: Fruquintinib 5 mg | Dose Expansion Phase, Cohort A: Fruquintinib 5 mg | Dose Expansion Phase, Cohort B: Fruquintinib 5 mg | Dose Expansion Phase, Cohort C: Fruquintinib 5 mg | Dose Expansion Phase, Cohort D: Fruquintinib 5 mg | Dose Expansion Phase, Cohort E: Fruquintinib 5 mg | Total
Number analyzed (Participants) | 7 | 7 | 6 | 41 | 40 | 14 | 14 | 129
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.08 (5.566) | 57.72 (12.712) | 68.91 (8.879) | 58.54 (10.182) | 56.94 (9.923) | 55.45 (13.443) | 50.86 (9.152) | 57.45 (10.672)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 3 | 21 | 24 | 14 | 14 | 86
  Male | 3 | 1 | 3 | 20 | 16 | 0 | 0 | 43
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 0 | 2 | 1 | 0 | 1 | 6
  Not Hispanic or Latino | 6 | 6 | 6 | 38 | 39 | 13 | 13 | 121
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 3 | 0 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 4 | 4 | 0 | 4 | 13
  White | 7 | 6 | 6 | 33 | 33 | 13 | 9 | 107
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 3 | 0 | 1 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Dose Escalation Phase: Number of Participants With Dose-limiting Toxicities (DLTs)
Description: Dose-limiting toxicity was defined as: Any Grade 4 non-hematologic toxicity; Any Grade 3 non-hematologic toxicity related to study drug except for nausea/vomiting, diarrhea, constipation, hypertension, and electrolyte imbalances downgraded within 3-days with appropriate supportive treatment; Grade 4 neutropenia lasting >3 days; Grade 3 febrile neutropenia (absolute neutrophil count [ANC] <1.0*10^9 per liter [/L] with a single temperature of greater than (>) 38.3 degree centigrade (°C) or a sustained temperature of greater than or equal to (>=) 38°C for more than 1 hour); Grade 4 thrombocytopenia or Grade 3 thrombocytopenia associated with bleeding; Dose interruption for >14 days due to toxicity.
Time Frame: Cycle 1 (cycle length equal to [=] 28 days)
Population: The DLT evaluable set comprised all participants who were evaluable for DLT assessment. As planned, this outcome measure (OM) was assessed in Dose Escalation Phase only.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation Phase: Fruquintinib 3 mg | Dose Escalation Phase: Fruquintinib 5 mg
Number analyzed (Participants) | 7 | 7
Participants | 1 | 0

2. Primary Outcome: Dose Escalation Phase: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious TEAEs
Description: TEAEs were defined as AEs that started or worsened in severity on or after the first dose of study medication and no later than 37 days after the date of last study treatment. A serious adverse event (SAE) was any AE that had any of the following characteristics: Fatal (that was, the AE actually caused or led to death, except for deaths caused by the progress of disease); Life threatening (that was, AE, in view of the investigator, places participant at immediate risk of death); Required or prolonged inpatient hospitalization (excluding emergency or outpatient treatment); Resulted in persistent or significant disability/incapacity (that was, the AE resulted in substantial disruption of the participant's ability to conduct normal life functions).
Time Frame: From first dose of study drug up to 37 days after last dose of study drug (i.e., up to 29 months)
Population: The SAS included all participants who received at least 1 dose of the study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation Phase: Fruquintinib 3 mg | Dose Escalation Phase: Fruquintinib 5 mg
Number analyzed (Participants) | 7 | 7
Participants
  Participants with TEAEs | 7 | 7
  Participants with serious TEAEs | 3 | 2

3. Primary Outcome: Dose Expansion Phase: Progression Free Survival (PFS) Rate
Description: PFS was defined as time from date of first dosing until date of an objective disease progression (PD) as defined by Response Evaluation Criteria in Solid Tumors (RECIST) Version (v) 1.1 or death due to any cause, whichever comes first. PFS was determined using all data until last evaluable visit prior to or on date of: (i) radiographic PD per RECIST v1.1; (ii) withdrawal of consent to obtain additional scans on study; or (iii) initiation of subsequent anticancer therapy other than study drugs, whichever was earlier. PFS rate was defined as probability of being disease progression free at selected timepoints such as 16 weeks and was calculated using Brookmeyer-Crowley method based on PFS events observed up to 29 months. PD:at least 20 percent (%) increase in sum of diameters of target lesions, taking as reference smallest sum on study, including baseline; an absolute increase of at least 5 millimeter (mm) in sum of diameters of target lesions; and appearance of one or more new lesions.
Time Frame: From the first dose of study drug to disease progression, or death, whichever occurred first (i.e., up to 29 months)
Population: The SAS included all participants who received at least 1 dose of the study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dose Expansion Phase, Cohort A: Fruquintinib 5 mg | Dose Expansion Phase, Cohort B: Fruquintinib 5 mg | Dose Expansion Phase, Cohort C: Fruquintinib 5 mg | Dose Expansion Phase, Cohort D: Fruquintinib 5 mg | Dose Expansion Phase, Cohort E: Fruquintinib 5 mg
Number analyzed (Participants) | 6 | 41 | 40 | 14 | 14
percentage of participants | 53.33 [4.68 to 100.00] | 61.04 [45.59 to 76.49] | 55.64 [39.87 to 71.41] | 29.30 [1.91 to 56.70] | 38.46 [12.02 to 64.91]

4. Secondary Outcome: Dose Escalation and Expansion Phase: Maximum Observed Plasma Concentration (Cmax) of Fruquintinib
Description: Cmax of fruquintinib was reported.
Time Frame: Dose Escalation and Cohort A of Expansion Phases: Predose, 1, 2, 4, 8, 24 hours post-dose on Days 1, 14, and 21 of Cycle 1; Cohorts B, C, D, E of Expansion Phase: Predose, 1, 2, 4, 8, 24 hours post-dose on Days 1 and 14 of Cycle 1 (Cycle 1 length=28 days)
Population: Pharmacokinetic (PK) evaluable population included all participants who received at least 1 dose of the study drug and had a sufficient PK profile to derive at least 1 PK parameter. Here, "number analyzed" signifies participants who were evaluable at specified timepoints. As per planned analysis, PK data were collected and reported for all cohorts at Cycle 1 Days 1 and 14; and for the Dose Escalation Phase and Cohort A of Expansion Phase at Cycle 1 Day 21 only.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Dose Escalation Phase: Fruquintinib 3 mg | Dose Escalation Phase: Fruquintinib 5 mg | Dose Expansion Phase, Cohort A: Fruquintinib 5 mg | Dose Expansion Phase, Cohort B: Fruquintinib 5 mg | Dose Expansion Phase, Cohort C: Fruquintinib 5 mg | Dose Expansion Phase, Cohort D: Fruquintinib 5 mg | Dose Expansion Phase, Cohort E: Fruquintinib 5 mg
Number analyzed (Participants) | 7 | 7 | 6 | 41 | 40 | 14 | 14
nanogram per milliliter (ng/mL)
  Cycle 1 Day 1 | 52.2 (24.2) | 114 (27.5) | 96.0 (23.0) | 85.2 (32.1) | 89.0 (43.2) | 104 (37.0) | 105 (36.5)
  Cycle 1 Day 14: number analyzed (Participants) | 5 | 6 | 2 | 34 | 33 | 12 | 10
  Cycle 1 Day 14 | 198 (9.8) | 403 (33.7) | 336 (50.9) | 271 (26.5) | 293 (27.1) | 331 (36.1) | 352 (23.4)
  Cycle 1 Day 21: number analyzed (Participants) | 5 | 6 | 1 | 0 | 0 | 0 | 0
  Cycle 1 Day 21 | 205 (12.8) | 390 (19.1) | 238 (NA) — Geometric Coefficient of Variation was not calculated due to single participant. |  |  |  |

5. Secondary Outcome: Dose Escalation and Expansion Phase: Time to Reach Maximum Observed Plasma Concentration (Tmax) of Fruquintinib
Description: Tmax of fruquintinib over a dosing intervals were reported.
Time Frame: as for outcome 4
Population: PK evaluable population included all participants who received at least 1 dose of the study drug and had a sufficient PK profile to derive at least 1 PK parameter. Here, "number analyzed" signifies participants who were evaluable at specified timepoints. As per planned analysis, PK data were collected and reported for all cohorts at Cycle 1 Days 1 and 14; and for the Dose Escalation Phase and Cohort A of Expansion Phase at Cycle 1 Day 21 only.
Measure: Median (Full Range); unit: hours
Arm/Group | Dose Escalation Phase: Fruquintinib 3 mg | Dose Escalation Phase: Fruquintinib 5 mg | Dose Expansion Phase, Cohort A: Fruquintinib 5 mg | Dose Expansion Phase, Cohort B: Fruquintinib 5 mg | Dose Expansion Phase, Cohort C: Fruquintinib 5 mg | Dose Expansion Phase, Cohort D: Fruquintinib 5 mg | Dose Expansion Phase, Cohort E: Fruquintinib 5 mg
Number analyzed (Participants) | 7 | 7 | 6 | 41 | 40 | 14 | 14
hours
  Cycle 1 Day 1 | 2.07 [1.03 to 21.2] | 1.95 [0.917 to 25.0] | 1.96 [1.00 to 13.8] | 2.25 [0.917 to 23.8] | 2.04 [0.983 to 2.04] | 2.00 [1.00 to 18.4] | 2.01 [1.75 to 23.9]
  Cycle 1 Day 14: number analyzed (Participants) | 5 | 6 | 2 | 34 | 33 | 12 | 10
  Cycle 1 Day 14 | 1.03 [0.967 to 1.92] | 2.00 [1.97 to 7.05] | 1.52 [1.00 to 2.03] | 2.03 [0.00 to 26.1] | 2.00 [0.933 to 7.18] | 1.86 [0.917 to 7.00] | 1.84 [0.933 to 7.00]
  Cycle 1 Day 21: number analyzed (Participants) | 5 | 6 | 1 | 0 | 0 | 0 | 0
  Cycle 1 Day 21 | 1.83 [0.917 to 1.98] | 2.00 [1.88 to 4.08] | 1.00 [NA to NA] — Full Range (minimum-maximum) was not calculated due to single participant. |  |  |  |

6. Secondary Outcome: Dose Escalation and Expansion Phase: Minimum Observed Plasma Concentration (Cmin) of Fruquintinib
Description: Cmin of fruquintinib was reported.
Time Frame: Dose Escalation and Cohort A of Expansion Phases: Predose, 1, 2, 4, 8, 24 hours post-dose on Days 14, and 21 of Cycle 1; Cohorts B, C, D, E of Expansion Phase: Predose, 1, 2, 4, 8, 24 hours post-dose on Day 14 of Cycle 1 (Cycle 1 length=28 days)
Population: PK evaluable population: all participants who received at least 1 dose of study drug and had a sufficient PK profile to derive at least 1 PK parameter. "Overall number of participants analyzed" signifies participants evaluable for this OM; "number analyzed" signifies participants evaluable at specified timepoints. As per planned analysis, PK data were collected and reported for all cohorts at Cycle 1 Day 14; and for Dose Escalation Phase and Cohort A of Expansion Phase at Cycle 1 Day 21 only.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Dose Escalation Phase: Fruquintinib 3 mg | Dose Escalation Phase: Fruquintinib 5 mg | Dose Expansion Phase, Cohort A: Fruquintinib 5 mg | Dose Expansion Phase, Cohort B: Fruquintinib 5 mg | Dose Expansion Phase, Cohort C: Fruquintinib 5 mg | Dose Expansion Phase, Cohort D: Fruquintinib 5 mg | Dose Expansion Phase, Cohort E: Fruquintinib 5 mg
Number analyzed (Participants) | 5 | 6 | 2 | 34 | 33 | 12 | 10
ng/mL
  Cycle 1 Day 14 | 138 (28.3) | 281 (101) | 251 (114) | 193 (57.3) | 204 (63.2) | 227 (98.4) | 249 (72.1)
  Cycle 1 Day 21: number analyzed (Participants) | 5 | 6 | 1 | 0 | 0 | 0 | 0
  Cycle 1 Day 21 | 140 (27.0) | 283 (81.0) | 182 (NA) — Standard Deviation was not calculated due to single participant. |  |  |  |

7. Secondary Outcome: Dose Escalation and Expansion Phase: Time to Reach Minimum Observed Plasma Concentration (Tmin) of Fruquintinib
Description: Tmin of fruquintinib was reported.
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Median (Full Range); unit: hours
Arm/Group | Dose Escalation Phase: Fruquintinib 3 mg | Dose Escalation Phase: Fruquintinib 5 mg | Dose Expansion Phase, Cohort A: Fruquintinib 5 mg | Dose Expansion Phase, Cohort B: Fruquintinib 5 mg | Dose Expansion Phase, Cohort C: Fruquintinib 5 mg | Dose Expansion Phase, Cohort D: Fruquintinib 5 mg | Dose Expansion Phase, Cohort E: Fruquintinib 5 mg
Number analyzed (Participants) | 5 | 6 | 2 | 34 | 33 | 12 | 10
hours
  Cycle 1 Day 14 | 0.00 [0.00 to 7.00] | 0.508 [0.00 to 27.8] | 3.57 [0.00 to 7.13] | 0.00 [0.00 to 25.6] | 0.00 [0.00 to 28.2] | 0.00 [0.00 to 23.9] | 0.458 [0.00 to 22.0]
  Cycle 1 Day 21: number analyzed (Participants) | 5 | 6 | 1 | 0 | 0 | 0 | 0
  Cycle 1 Day 21 | 7.00 [0.00 to 25.6] | 3.54 [0.00 to 24.9] | 7.00 [NA to NA] — Full Range (minimum-maximum) was not calculated due to single participant. |  |  |  |

8. Secondary Outcome: Dose Escalation and Expansion Phase: Area Under the Plasma Concentration-time Curve From Time 0 to 24 Hours (AUC0-24) of Fruquintinib
Description: AUC0-24 of fruquintinib was reported.
Time Frame: as for outcome 4
Population: PK evaluable population:all participants who received at least 1 dose of study drug and had a sufficient PK profile to derive at least 1 PK parameter. "Overall number of participants analyzed" signifies participants evaluable for this OM; "number analyzed" signifies participants evaluable at specified timepoints. As per planned analysis, PK data were collected and reported for all cohorts at Cycle 1 Days 1 and 14; and for Dose Escalation Phase, Cohort A of Expansion Phase at Cycle 1 Day 21 only.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanogram per millimeter (h*ng/mL)
Arm/Group | Dose Escalation Phase: Fruquintinib 3 mg | Dose Escalation Phase: Fruquintinib 5 mg | Dose Expansion Phase, Cohort A: Fruquintinib 5 mg | Dose Expansion Phase, Cohort B: Fruquintinib 5 mg | Dose Expansion Phase, Cohort C: Fruquintinib 5 mg | Dose Expansion Phase, Cohort D: Fruquintinib 5 mg | Dose Expansion Phase, Cohort E: Fruquintinib 5 mg
Number analyzed (Participants) | 6 | 7 | 3 | 34 | 33 | 12 | 10
hour*nanogram per millimeter (h*ng/mL)
  Cycle 1 Day 1: number analyzed (Participants) | 6 | 7 | 3 | 33 | 33 | 11 | 8
  Cycle 1 Day 1 | 912 (21.5) | 2010 (19.2) | 1340 (25.6) | 1384 (39.0) | 1550 (46.5) | 1821 (31.5) | 1739 (39.8)
  Cycle 1 Day 14: number analyzed (Participants) | 5 | 6 | 2 | 34 | 33 | 12 | 10
  Cycle 1 Day 14 | 3694 (17.1) | 8249 (35.2) | 6507 (53.7) | 5338 (28.9) | 5833 (27.3) | 6135 (40.1) | 6957 (25.1)
  Cycle 1 Day 21: number analyzed (Participants) | 5 | 6 | 1 | 0 | 0 | 0 | 0
  Cycle 1 Day 21 | 3731 (22.5) | 7740 (26.7) | 4995 (NA) — Geometric Coefficient of Variation was not calculated due to single participant. |  |  |  |

9. Secondary Outcome: Dose Escalation and Expansion Phase: Apparent Clearance at Steady State (CL/Fss) of Fruquintinib
Description: CL/Fss was calculated as Dose/AUC0-t. As planned, CL/Fss was assessed at Cycle 1 Days 14 and 21 after multiple dose administration in Dose Escalation Phase and Cohort A of Dose Expansion Phase; and at Cycle 1 Day 14 for Cohort B, C, D, E of Expansion Phase.
Time Frame: as for outcome 6
Population: PK evaluable population:all participants who received at least 1 dose of the study drug and had a sufficient PK profile to derive at least 1 PK parameter. "Overall number of participants analyzed" signifies participants evaluable for this OM; "number analyzed" signifies participants evaluable at specified timepoints. As per planned analysis, PK data were collected and reported for all cohorts at Cycle 1 Day 14; and for Dose Escalation Phase and Cohort A of Expansion Phase at Cycle 1 Day 21 only.
Measure: Mean (Standard Deviation); unit: milliliter per minute (mL/min)
Arm/Group | Dose Escalation Phase: Fruquintinib 3 mg | Dose Escalation Phase: Fruquintinib 5 mg | Dose Expansion Phase, Cohort A: Fruquintinib 5 mg | Dose Expansion Phase, Cohort B: Fruquintinib 5 mg | Dose Expansion Phase, Cohort C: Fruquintinib 5 mg | Dose Expansion Phase, Cohort D: Fruquintinib 5 mg | Dose Expansion Phase, Cohort E: Fruquintinib 5 mg
Number analyzed (Participants) | 4 | 6 | 2 | 34 | 33 | 12 | 10
milliliter per minute (mL/min)
  Cycle 1 Day 14 | 14.4 (2.90) | 11.1 (4.04) | 14.1 (7.31) | 16.3 (5.16) | 14.8 (3.92) | 14.7 (7.18) | 12.3 (2.80)
  Cycle 1 Day 21: number analyzed (Participants) | 4 | 6 | 1 | 0 | 0 | 0 | 0
  Cycle 1 Day 21 | 14.1 (3.07) | 11.3 (2.83) | 17.5 (NA) — Standard Deviation was not calculated due to single participant. |  |  |  |

10. Secondary Outcome: Dose Escalation and Expansion Phase: Accumulation Ratio Based on Cmax of Fruquintinib
Description: Accumulation ratio based on Cmax for Cycle 1 Day 14 was calculated as Day 14 Cmax /Day 1 Cmax and for Cycle 1 Day 21 was calculated as Day 21 Cmax /Day 1 Cmax. Accumulation ratio based on Cmax of fruquintinib was reported.
Time Frame: Dose Escalation and Cohort A of Expansion Phases: Predose, 1, 2, 4, 8, 24 hours post-dose on Days 14 and 21 of Cycle 1; Cohorts B, C, D, E of Expansion Phase: Predose, 1, 2, 4, 8, 24 hours post-dose on Day 14 of Cycle 1 (Cycle 1 length=28 days)
Population: PK evaluable population: all participants who received at least 1 dose of study drug and had a sufficient PK profile to derive at least 1 PK parameter. Here, "overall number of participants analyzed" signifies participants evaluable for this OM; "number analyzed" signifies participants evaluable at specified timepoints. As per planned analysis, PK data were collected and reported for all cohorts at Cycle 1 Day 14; and for Dose Escalation Phase, Cohort A of Expansion Phase at Cycle 1 Day 21 only.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Dose Escalation Phase: Fruquintinib 3 mg | Dose Escalation Phase: Fruquintinib 5 mg | Dose Expansion Phase, Cohort A: Fruquintinib 5 mg | Dose Expansion Phase, Cohort B: Fruquintinib 5 mg | Dose Expansion Phase, Cohort C: Fruquintinib 5 mg | Dose Expansion Phase, Cohort D: Fruquintinib 5 mg | Dose Expansion Phase, Cohort E: Fruquintinib 5 mg
Number analyzed (Participants) | 5 | 6 | 2 | 34 | 33 | 12 | 10
ratio
  Cycle 1 Day 14 | 4.06 (1.42) | 3.66 (1.42) | 3.57 (0.232) | 3.32 (1.21) | 3.44 (1.36) | 3.22 (1.38) | 3.40 (0.963)
  Cycle 1 Day 21: number analyzed (Participants) | 5 | 6 | 1 | 0 | 0 | 0 | 0
  Cycle 1 Day 21 | 4.22 (1.45) | 3.47 (1.22) | 3.40 (NA) — Standard Deviation was not calculated due to single participant. |  |  |  |

11. Secondary Outcome: Dose Escalation and Expansion Phase: Accumulation Ratio Based on AUC0-24 Hours of Fruquintinib
Description: Accumulation ratio for Cycle 1 Day 14 was calculated as AUC0-24 at Day 14 divided by AUC0-24h at Day 1, and for Cycle 1 Day 21 was calculated as AUC0-24 at Day 21 divided by AUC0-24 at Day 1. Accumulation ratio based on AUC0-24 of fruquintinib was reported.
Time Frame: as for outcome 10
Population: PK evaluable population included all participants who received at least 1 dose of the study drug and had a sufficient PK profile to derive at least 1 PK parameter. Here, "overall number of participants analyzed" signifies participants who were evaluable for this OM. As per planned analysis, PK data were collected and reported for all cohorts at Cycle 1 Day 14; and for Dose Escalation Phase and Cohort A of Expansion Phase at Cycle 1 Day 21 only.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Dose Escalation Phase: Fruquintinib 3 mg | Dose Escalation Phase: Fruquintinib 5 mg | Dose Expansion Phase, Cohort A: Fruquintinib 5 mg | Dose Expansion Phase, Cohort B: Fruquintinib 5 mg | Dose Expansion Phase, Cohort C: Fruquintinib 5 mg | Dose Expansion Phase, Cohort D: Fruquintinib 5 mg | Dose Expansion Phase, Cohort E: Fruquintinib 5 mg
Number analyzed (Participants) | 5 | 6 | 1 | 28 | 28 | 9 | 6
ratio
  Cycle 1 Day 14 | 4.24 (1.21) | 4.19 (1.19) | 4.04 (NA) — Standard Deviation was not calculated due to single participant. | 3.87 (1.22) | 4.38 (3.08) | 3.73 (1.51) | 4.37 (1.70)
  Cycle 1 Day 21: number analyzed (Participants) | 5 | 6 | 1 | 0 | 0 | 0 | 0
  Cycle 1 Day 21 | 4.36 (1.53) | 3.90 (0.964) | 4.43 (NA) — Standard Deviation was not calculated due to single participant. |  |  |  |

12. Secondary Outcome: Dose Escalation and Expansion Phase: Objective Response Rate (ORR)
Description: ORR was defined as the percentage of participants with objective complete response (CR) or partial response (PR) response per RECIST version 1.1. As per RECIST 1.1; CR was defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR was defined at least a 30 percent (%) decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters.
Time Frame: From the first dose of study drug until first documentation of best overall response (i.e., up to 29 months)
Population: The Efficacy Analysis Set included all participants who received at least 1 dose of fruquintinib, had a measurable lesion (target lesions >=10 mm) at the baseline tumor assessment, and either: 1) had at least 1 postbaseline tumor assessment; or 2) did not have post-dose tumor assessment but had clinical progression as noted by the Investigator; or died due to disease progression before their first postbaseline tumor scan.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dose Escalation Phase: Fruquintinib 3 mg | Dose Escalation Phase: Fruquintinib 5 mg | Dose Expansion Phase, Cohort A: Fruquintinib 5 mg | Dose Expansion Phase, Cohort B: Fruquintinib 5 mg | Dose Expansion Phase, Cohort C: Fruquintinib 5 mg | Dose Expansion Phase, Cohort D: Fruquintinib 5 mg | Dose Expansion Phase, Cohort E: Fruquintinib 5 mg
Number analyzed (Participants) | 6 | 7 | 6 | 41 | 39 | 10 | 13
percentage of participants | 16.7 [0.42 to 64.12] | 14.3 [0.36 to 57.87] | 0.0 [0.00 to 45.93] | 2.4 [0.06 to 12.86] | 5.1 [0.63 to 17.32] | 0.0 [0.00 to 30.85] | 0.0 [0.00 to 24.71]

13. Secondary Outcome: Dose Escalation and Expansion Phase: Disease Control Rate (DCR)
Description: DCR was defined as the percentage of participants with a best overall response (BOR) of confirmed CR, confirmed PR or stable disease (SD) (for 7 weeks) per RECIST version 1.1. As per RECIST 1.1; CR was defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR was defined at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters. SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study [this might include the baseline sum]).
Time Frame: From the first dose of study drug until first documentation of best overall response (i.e., up to 29 months)
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dose Escalation Phase: Fruquintinib 3 mg | Dose Escalation Phase: Fruquintinib 5 mg | Dose Expansion Phase, Cohort A: Fruquintinib 5 mg | Dose Expansion Phase, Cohort B: Fruquintinib 5 mg | Dose Expansion Phase, Cohort C: Fruquintinib 5 mg | Dose Expansion Phase, Cohort D: Fruquintinib 5 mg | Dose Expansion Phase, Cohort E: Fruquintinib 5 mg
Number analyzed (Participants) | 6 | 7 | 6 | 41 | 39 | 10 | 13
percentage of participants | 66.7 [22.28 to 95.67] | 71.4 [29.04 to 96.33] | 66.7 [22.28 to 95.67] | 68.3 [51.91 to 81.92] | 59.0 [42.10 to 74.43] | 60.0 [26.24 to 87.84] | 38.5 [13.86 to 68.42]

14. Secondary Outcome: Dose Escalation and Expansion Phase: Duration of Response (DoR)
Description: DoR was defined as the time (in months) from the date of the first objective response (CR or PR) until the date of the documented progression or of death, whichever comes first. DoR was only analyzed for participants whose best overall response (BOR) was either CR or PR. As per RECIST 1.1; CR was defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR was defined at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters. PD was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this might include the baseline sum). DoR was calculated using the Kaplan-Meier method.
Time Frame: From the date of the first objective response (CR or PR) until the date of the documented disease progression or of death, whichever comes first (i.e., up to 29 months)
Population: Efficacy Analysis Set was used for analysis. Here, "Overall number of participants analyzed" signifies participants who had CR or PR; & '0' in 'overall number of participants analyzed represents that DOR could only be analyzed in participants who achieved a response i.e., CR or PR. As no participant in the dose expansion cohorts A, D and E achieved any response, no DOR is available.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Dose Escalation Phase: Fruquintinib 3 mg | Dose Escalation Phase: Fruquintinib 5 mg | Dose Expansion Phase, Cohort A: Fruquintinib 5 mg | Dose Expansion Phase, Cohort B: Fruquintinib 5 mg | Dose Expansion Phase, Cohort C: Fruquintinib 5 mg | Dose Expansion Phase, Cohort D: Fruquintinib 5 mg | Dose Expansion Phase, Cohort E: Fruquintinib 5 mg
Number analyzed (Participants) | 1 | 1 | 0 | 1 | 2 | 0 | 0
months | 7.56 [NA to NA] — 95% Confidence Interval (CI) was not determined due to insufficient numbers of participants with events. | NA [NA to NA] — Median and 95% CI was not determined due to insufficient numbers of participants with events. |  | 4.04 [NA to NA] — 95% CI was not determined due to insufficient numbers of participants with events. | NA [5.65 to NA] — Median and upper limit of 95% CI was not determined due to insufficient numbers of participants with events. |  |

15. Secondary Outcome: Dose Escalation and Expansion Phase: Progression Free Survival (PFS)
Description: PFS was defined as the time (in months) from date of first dosing until the date of an objective disease progression as per RECIST version 1.1 or death due to any cause, whichever comes first. PFS was determined using all the assessment data up until the last evaluable visit prior to or on the date of (i) disease progression as defined by RECIST version 1.1 or death; or (ii) withdrawal of consent; or (iii) receiving subsequent anti-cancer therapy, whichever is earlier. Disease progression was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this might include the baseline sum). PFS was calculated using the Kaplan-Meier method.
Time Frame: From date of first dose until the date of an objective disease progression or death due to any cause, whichever comes first (i.e., up to 29 months)
Population: The SAS included all participants who received at least 1 dose of the study drug.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Dose Escalation Phase: Fruquintinib 3 mg | Dose Escalation Phase: Fruquintinib 5 mg | Dose Expansion Phase, Cohort A: Fruquintinib 5 mg | Dose Expansion Phase, Cohort B: Fruquintinib 5 mg | Dose Expansion Phase, Cohort C: Fruquintinib 5 mg | Dose Expansion Phase, Cohort D: Fruquintinib 5 mg | Dose Expansion Phase, Cohort E: Fruquintinib 5 mg
Number analyzed (Participants) | 7 | 7 | 6 | 41 | 40 | 14 | 14
months | 6.90 [0.56 to NA] — Upper limit of 95% CI was not determined due to insufficient numbers of participants with events. | NA [3.65 to NA] — Median and upper limit of 95% CI was not determined due to insufficient numbers of participants with events. | 5.49 [1.77 to NA] — Upper limit of 95% CI was not determined due to insufficient numbers of participants with events. | 4.67 [2.76 to 5.32] | 3.75 [2.00 to 5.49] | 2.43 [1.74 to 5.06] | 1.87 [1.15 to 3.94]

16. Secondary Outcome: Dose Escalation and Expansion Phase: Overall Survival (OS)
Description: OS was defined as the time interval (in months) between the first dose date and the date of death (any cause). OS was calculated using the Kaplan-Meier method.
Time Frame: From first dose date to the date of death (due to any cause) (i.e., up to 29 months)
Population: The SAS included all participants who received at least 1 dose of the study drug.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Dose Escalation Phase: Fruquintinib 3 mg | Dose Escalation Phase: Fruquintinib 5 mg | Dose Expansion Phase, Cohort A: Fruquintinib 5 mg | Dose Expansion Phase, Cohort B: Fruquintinib 5 mg | Dose Expansion Phase, Cohort C: Fruquintinib 5 mg | Dose Expansion Phase, Cohort D: Fruquintinib 5 mg | Dose Expansion Phase, Cohort E: Fruquintinib 5 mg
Number analyzed (Participants) | 7 | 7 | 6 | 41 | 40 | 14 | 14
months | 22.70 [0.56 to NA] — Upper limit of 95% CI was not determined due to insufficient numbers of participants with events. | 19.58 [6.05 to NA] — Upper limit of 95% CI was not determined due to insufficient numbers of participants with events. | 6.03 [4.24 to NA] — Upper limit of 95% CI was not determined due to insufficient numbers of participants with events. | 8.71 [6.57 to 11.47] | 10.64 [5.16 to 19.32] | 12.06 [6.21 to 13.24] | 8.74 [3.78 to 15.93]

17. Secondary Outcome: Dose Escalation and Expansion Phase: Percent Change From Baseline (PCFB) in Tumor Size
Description: Tumor size was estimated using data on sum of diameters of target lesion. Percentage change in tumor size from baseline was determined for participants with measurable disease at baseline and derived by the percentage change in the sum of the diameters of target lesions (TLs) compared to baseline. Baseline was defined as the last evaluable tumor assessment result obtained prior to the first administration of study medication.
Time Frame: Baseline up to 29 months
Population: Efficacy Analysis Set: all participants who received at least 1 dose of fruquintinib, had a measurable lesion (target lesions >=10 mm) at baseline tumor assessment and either: 1) had at least 1 postbaseline tumor assessment; or 2) did not have post-dose tumor assessment but had clinical progression as noted by Investigator; or died due to disease progression before first postbaseline tumor scan. Overall number of participants analyzed signifies participants evaluable for this OM.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Dose Escalation Phase: Fruquintinib 3 mg | Dose Escalation Phase: Fruquintinib 5 mg | Dose Expansion Phase, Cohort A: Fruquintinib 5 mg | Dose Expansion Phase, Cohort B: Fruquintinib 5 mg | Dose Expansion Phase, Cohort C: Fruquintinib 5 mg | Dose Expansion Phase, Cohort D: Fruquintinib 5 mg | Dose Expansion Phase, Cohort E: Fruquintinib 5 mg
Number analyzed (Participants) | 1 | 2 | 2 | 19 | 15 | 3 | 3
percent change | 5.41 (NA) — Standard Deviation was not calculated for singe participant. | -20.70 (16.485) | -12.92 (25.919) | 7.40 (23.713) | 19.23 (20.808) | -8.07 (8.574) | 9.82 (16.824)

18. Secondary Outcome: Dose Expansion Phase: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious TEAEs
Description: TEAEs were defined as AEs that started or worsened in severity on or after the first dose of study medication and no later than 37 days after the date of last study treatment. A SAE was any AE that had any of the following characteristics: Fatal (that was, the AE actually caused or led to death, except for deaths caused by the progress of disease); Life threatening (that was, AE, in view of the investigator, places participant at immediate risk of death); Required or prolonged inpatient hospitalization (excluding emergency or outpatient treatment); Resulted in persistent or significant disability/incapacity (that was, the AE resulted in substantial disruption of the participant's ability to conduct normal life functions).
Time Frame: From first dose of study drug up to 37 days after last dose of study drug (i.e., up to 29 months)
Population: The SAS included all participants who received at least 1 dose of the study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Expansion Phase, Cohort A: Fruquintinib 5 mg | Dose Expansion Phase, Cohort B: Fruquintinib 5 mg | Dose Expansion Phase, Cohort C: Fruquintinib 5 mg | Dose Expansion Phase, Cohort D: Fruquintinib 5 mg | Dose Expansion Phase, Cohort E: Fruquintinib 5 mg
Number analyzed (Participants) | 6 | 41 | 40 | 14 | 14
Participants
  Participants with TEAEs | 6 | 41 | 39 | 14 | 14
  Participants with serious TEAEs | 4 | 19 | 14 | 2 | 4

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to 37 days after last dose of study drug (i.e., up to 29 months)
Description: The SAS included all participants who received at least 1 dose of the study drug.
Arm/Group | Dose Escalation Phase: Fruquintinib 3 mg | Dose Escalation Phase: Fruquintinib 5 mg | Dose Expansion Phase, Cohort A: Fruquintinib 5 mg | Dose Expansion Phase, Cohort B: Fruquintinib 5 mg | Dose Expansion Phase, Cohort C: Fruquintinib 5 mg | Dose Expansion Phase, Cohort D: Fruquintinib 5 mg | Dose Expansion Phase, Cohort E: Fruquintinib 5 mg
All-Cause Mortality (participants affected / at risk) | 3/7 | 2/7 | 3/6 | 30/41 | 25/40 | 12/14 | 12/14
Serious Adverse Events (participants affected / at risk) | 3/7 | 2/7 | 4/6 | 19/41 | 14/40 | 2/14 | 4/14
Other Adverse Events (participants affected / at risk) | 7/7 | 7/7 | 6/6 | 41/41 | 39/40 | 14/14 | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Escalation Phase: Fruquintinib 3 mg (N=7) | Dose Escalation Phase: Fruquintinib 5 mg (N=7) | Dose Expansion Phase, Cohort A: Fruquintinib 5 mg (N=6) | Dose Expansion Phase, Cohort B: Fruquintinib 5 mg (N=41) | Dose Expansion Phase, Cohort C: Fruquintinib 5 mg (N=40) | Dose Expansion Phase, Cohort D: Fruquintinib 5 mg (N=14) | Dose Expansion Phase, Cohort E: Fruquintinib 5 mg (N=14)
Acquired oesophageal web (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Breast cellulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Osteomyelitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 2 | 1 | 0 | 0
Embolic stroke (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 1 | 1 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 3 | 3 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Gastric ulcer perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Cholecystitis infective (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Device related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Kidney infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Biliary obstruction (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Death (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Systemic inflammatory response syndrome (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Cognitive disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Escalation Phase: Fruquintinib 3 mg (N=7) | Dose Escalation Phase: Fruquintinib 5 mg (N=7) | Dose Expansion Phase, Cohort A: Fruquintinib 5 mg (N=6) | Dose Expansion Phase, Cohort B: Fruquintinib 5 mg (N=41) | Dose Expansion Phase, Cohort C: Fruquintinib 5 mg (N=40) | Dose Expansion Phase, Cohort D: Fruquintinib 5 mg (N=14) | Dose Expansion Phase, Cohort E: Fruquintinib 5 mg (N=14)
Diarrhoea (Gastrointestinal disorders) | 3 | 3 | 5 | 17 | 5 | 5 | 4
Nausea (Gastrointestinal disorders) | 4 | 4 | 1 | 11 | 6 | 7 | 7
Constipation (Gastrointestinal disorders) | 5 | 3 | 3 | 11 | 6 | 6 | 3
Abdominal pain (Gastrointestinal disorders) | 3 | 3 | 0 | 8 | 7 | 5 | 3
Vomiting (Gastrointestinal disorders) | 4 | 4 | 3 | 7 | 3 | 2 | 4
Stomatitis (Gastrointestinal disorders) | 2 | 2 | 1 | 8 | 3 | 4 | 3
Oral pain (Gastrointestinal disorders) | 0 | 1 | 1 | 2 | 3 | 6 | 2
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1 | 5 | 0 | 3 | 1
Dyspepsia (Gastrointestinal disorders) | 2 | 3 | 1 | 3 | 0 | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 2 | 1 | 3 | 0 | 3 | 1
Oral dysaesthesia (Gastrointestinal disorders) | 0 | 2 | 2 | 2 | 1 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 2 | 2 | 0 | 2 | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 3 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 2 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 3 | 0 | 1 | 0
Glossodynia (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Acquired oesophageal web (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Anal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Eructation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Faeces pale (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lip swelling (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 2 | 1 | 11 | 11 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 10 | 9 | 1 | 3
Weight decreased (Investigations) | 2 | 4 | 0 | 9 | 4 | 1 | 3
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 6 | 9 | 2 | 1
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 7 | 9 | 0 | 1
International normalised ratio increased (Investigations) | 1 | 0 | 0 | 9 | 5 | 0 | 1
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 7 | 8 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 1 | 3 | 9 | 0 | 0
Platelet count decreased (Investigations) | 0 | 1 | 0 | 6 | 3 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 4 | 4 | 0 | 1
Blood cholesterol increased (Investigations) | 0 | 0 | 0 | 4 | 3 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 4 | 1 | 0 | 2
White blood cell count decreased (Investigations) | 0 | 1 | 0 | 3 | 2 | 0 | 1
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 1 | 3 | 0 | 2
Blood thyroid stimulating hormone increased (Investigations) | 0 | 1 | 0 | 1 | 1 | 0 | 1
Ejection fraction decreased (Investigations) | 0 | 0 | 0 | 1 | 2 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 3 | 0 | 0 | 0
Haemoglobin increased (Investigations) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Blood thyroid stimulating hormone decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Protein total decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Troponin I increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 2 | 3 | 5 | 20 | 29 | 9 | 6
Hypotension (Vascular disorders) | 0 | 0 | 0 | 3 | 2 | 0 | 3
Flushing (Vascular disorders) | 0 | 1 | 0 | 2 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Haemorrhage (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lymphoedema (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vasculitis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 4 | 2 | 14 | 10 | 4 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 11 | 10 | 1 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 8 | 11 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 6 | 9 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 6 | 3 | 1 | 2
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 6 | 3 | 1 | 2
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 3 | 2 | 1 | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 5 | 2 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 3 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 3 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 2 | 0 | 0
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0 | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 0
Increased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1 | 7 | 8 | 6 | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 2 | 13 | 5 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 4 | 6 | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 3 | 3 | 2 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 1 | 2 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 2 | 1 | 1 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 3 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 3 | 0 | 2 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 2 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Jaw clicking (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 1 | 3 | 2 | 22 | 12 | 8 | 5
Pyrexia (General disorders) | 1 | 1 | 0 | 2 | 4 | 1 | 1
Oedema peripheral (General disorders) | 1 | 1 | 0 | 3 | 2 | 1 | 0
Non-cardiac chest pain (General disorders) | 2 | 0 | 0 | 1 | 1 | 0 | 2
Gait disturbance (General disorders) | 0 | 0 | 0 | 1 | 2 | 2 | 0
Influenza like illness (General disorders) | 1 | 0 | 0 | 3 | 0 | 0 | 1
Chills (General disorders) | 1 | 0 | 0 | 2 | 1 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 2 | 0 | 1 | 0
Chest discomfort (General disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 0
Axillary pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Device related thrombosis (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Generalised oedema (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tenderness (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 4 | 13 | 10 | 5 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 1 | 7 | 2 | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 3 | 5 | 1 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2 | 2 | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1 | 1 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 2 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 2 | 0 | 0
Bronchostenosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Laryngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 4 | 2 | 11 | 6 | 5 | 7
Dizziness (Nervous system disorders) | 2 | 1 | 3 | 4 | 2 | 2 | 1
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 3 | 3 | 2 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0
Dysarthria (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Tremor (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Burning sensation (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lethargy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Speech disorder (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Taste disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Proteinuria (Renal and urinary disorders) | 2 | 4 | 2 | 20 | 16 | 5 | 3
Haematuria (Renal and urinary disorders) | 0 | 2 | 2 | 4 | 2 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 1 | 0 | 1 | 1 | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 12 | 9 | 4 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 3 | 2 | 0 | 3
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 3
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 3 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rosacea (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Skin disorder (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 8 | 3 | 4 | 3
Upper respiratory tract infection (Infections and infestations) | 2 | 1 | 1 | 3 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 1 | 1 | 0 | 0 | 0
Candida infection (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Escherichia urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Localised infection (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Fungal foot infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gingivitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Otitis externa (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pyuria (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rash pustular (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Wound infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 1 | 2 | 1 | 7 | 11 | 6 | 4
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 0 | 1 | 2 | 2 | 2
Anxiety (Psychiatric disorders) | 2 | 1 | 1 | 1 | 1 | 2 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 0 | 6 | 2 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1 | 0 | 3 | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 1 | 0 | 3 | 0 | 0 | 0
Hallucination (Psychiatric disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 0 | 1 | 4 | 3 | 2 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 1 | 0 | 0 | 0
Vascular access complication (Injury, poisoning and procedural complications) | 1 | 1 | 1 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal wall wound (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Eye injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 4 | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Atrial flutter (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Left ventricular dysfunction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 6 | 4 | 1 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1 | 3 | 2 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 2 | 0 | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Vulvovaginal pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Brain neoplasm benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin neoplasm bleeding (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blindness unilateral (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Eye haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Contrast media allergy (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Seasonal allergy (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2020-01-09): https://cdn.clinicaltrials.gov/large-docs/78/NCT03251378/Prot_000.pdf
  • Statistical Analysis Plan (2022-02-18): https://cdn.clinicaltrials.gov/large-docs/78/NCT03251378/SAP_001.pdf